CLINICAL TRIAL: NCT03929549
Title: Preliminary Evaluation of a Remotely Controlled Mandibular Positioner to Predict Failure of Maxillomandibular Advancement Surgery for Obstructive Sleep Apnea
Brief Title: Preliminary Evaluation of a RCMP to Predict Failure of Maxillomandibular Advancement Surgery for OSA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Sharon Aronovich, Clinical Assistant Professor of Dentistry, Department of Oral and Maxillofacial Surgery, School of Dentistry and Assistant Professor of Oral Surgery, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: HUM00143739; M-ROSA trial (Other: University of Michigan)
Record Dates: First submitted 2019-04-24; First posted 2019-04-29 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Obstructive Sleep Apnea; Maxillomandibular Advancement Surgery
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- RCMP titration (Experimental): Remotely Controlled Mandibular Positioner
  Interventions: Device: RCMP titration

INTERVENTIONS:
Device: RCMP titration — An overnight titration polysomnogram with gradual mandibular protrusion and assessment of polysomnographic parameters (i.e. AHI, oxygen saturation, etc.) at various magnitudes of protrusion.
  Other Names: Remotely Controlled Mandibular Positioner

SUMMARY:
Maxillomandibular advancement (MMA) surgery, one of the most successful surgical procedures for the treatment of obstructive sleep apnea (OSA), is predominantly used to manage patients with moderate to severe OSA. However, limiting factors include incomplete response in some cases, unfavorable facial changes as a result of large advancements, and risk of malocclusion or malunion.

This study will be done to determine predictors of success with MMA surgery in patients with moderate to severe OSA. Studies have already shown the value of a remote controlled mandibular positioner (RCMP) device to identify the correct level of therapeutic protrusion needed with oral appliance therapy. Moreover, some patients experience a dose dependent improvement in sleep parameters based on the degree of protrusion during the titration study. Use of RCMP as a means to identify potential candidates for MMA, may help customize treatment options for patients with OSA by providing predictive value.

DETAILED DESCRIPTION:
The use of a remotely controlled mandibular protrusion (RCMP) device allows for customization of treatment by titrating the extent of mandibular protrusion during a polysomnogram. Use of the RCMP device has a high degree of positive and negative predictive value in determining the effectiveness and degree (effective target protrusive position) of mandibular advancement need with oral appliance therapy (Remmers, 2013). Preliminary data from 4 patients (Hoekena 2006) indicates that patients with a significant response to oral appliance therapy (>50% reduction in AHI) may have a better response to MMA. This study will determine the efficacy of MMA in patients with moderate to severe OSA, and determine if the RCMP titration can predict success or failure with MMA for treatment of OSA.

Patients will undergo detailed history and physical examination by Oral & Maxillofacial Surgery. Those patients found to be potential candidates for jaw advancement (MMA) surgery will be recruited to enroll in the study. Once consented and enrolled, study participants will undergo a titration study using a remote controlled mandibular positioner (RCMP titration study) to evaluate changes in polysomnographic parameters (i.e. Apnea-hypopnea index and oxygen saturation) with mandibular protrusion. Patients will then undergo maxillomandibular advancement surgery (MMA surgery). During MMA surgery, a standard 10 mm advancement of the upper and lower jaw is performed. Slight modifications may be made to the degree of advancement in order to achieve acceptable facial esthetics. Data from the RCMP titration study will not affect how the MMA surgery is performed. After surgery, participants will have a follow-up polysomnogram four to eight months post-operatively to assess for treatment response and compared this to the predicted response based on the RCMP titration study.

ELIGIBILITY:
Inclusion Criteria:

AHI ≥ 15/hour

30-65 years of age

BMI 25-34.9

Ideal operative candidate

Unable or unwilling to use PAP

Exclusion Criteria:

BMI ≥ 35

younger than 30 or older than 65 years of age

pregnancy

Central sleep apnea (CSA) on baseline polysomnogram

Chronic opioid use

Active TMJ Disorders

Inability to protrude the mandible beyond 5 mm

Inability to follow-up after surgery

Dental disorders including loose teeth or advanced periodontal disease

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-08-12 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Primary outcome variable: Change in AHI (pre-post) with MMA surgery | baseline (pre-operative), post surgery (6 months)
  Secondary outcome variable: Failure of MMA surgery defined as AHI ≥ 15/hour
Primary predictor variable: Change in AHI, from baseline to maximal therapeutic protrusion, with RCMP study | baseline (pre-operative), post surgery (6 months)
  age, sex, BMI, AHI, retrognathia, airway collapse on forced inspiration, AHI reduction on RCMP titration and magnitude of advancement.

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Aronovich, DMD, Principal Investigator — University of Michigan
Locations (1):
- Michigan Medicine Oral and Maxillofacial Surgery, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: Yes
We will share deidentified individual patient data which supports the results reported in research publications. The data will be published as supplemental files with the original publication.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Upon publication (Deidentified individual patient data may be published as supplemental files to an original research paper)
Access Criteria: Deidentified individual patient data shared with a published paper will be published as supplemental files with the original publication